CLINICAL TRIAL: NCT06723938
Title: Phenotypic and Genotypic Characterisation of a Large, Multicentre Italian Cohort of 46, XY DSD Patients
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: DSDPed
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: 46, XY DSD
Keywords: 46 XY DSD
MeSH Terms: conditions — Disorder of Sex Development, 46,XY

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Observational exploratory study of a cohort of pediatric and adolescent patients diagnosed with DSD karyotype 46,XY, a rare congenital clinical condition characterized by a disharmonic development between chromosomal sex, gonadal sex and/or phenotypic sex.

DETAILED DESCRIPTION:
Observational, retro-prospective, exploratory, multicentre study coordinate by the IRCCS Azienda Ospedaliero-Universitaria of Bologna, Italy.

The study consists of the collection and analysis of clinical, biochemical, instrumental and genetic data on pediatric and adolescent patients referred to partecipating centres in a given period with a diagnosis of 46,XY Disorders of Sex Development (DSD).

The primary aim of the study is to assess the number of 46,XY DSD patients referred to partecipating centres, describing the phenotypic, hormonal and genetic characterisation.

The secondary aims are to assess the correlation between molecular diagnosis and EMS/EGS score (External Masculinization Score ed ExternalGenital Score) and to evaluate the diagnostic rate over the reporting period.

ELIGIBILITY:
Inclusion Criteria:

* Karyotype 46,XY DSD;
* Genital ambiguity signs assessed on the basis of clinical phenotype and EMS/EGS for karyotype 46,XY DSD;
* Age < 18 years at diagnosis of 46,XY DSD;
* Patients referred to the IRCCS Azienda Ospedaliero-Universitaria di Bologna since 01/01/1991 or to other participating centres since 01/01/2000;
* Obtaining informed consent from patients or from parents/legal guardian of pediatric patients.

Exclusion Criteria:

• None.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged < 18 years at diagnosis of 46,XY DSD who referred to the IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy, since 01/01/1991 or to other participating italian centres since 01/01/2000.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of 46,XY DSD patients | 4 years after the start of enrollment
  number of 46,XY DSD patients referred to partecipating centres during the reporting period
Sex | at baseline
  sex assigned at birth, and current sex (M/F)
EMS/EGS (External Masculinization Score ed ExternalGenital Score) | at baseline
  presence/absence of micropenis, bifid scrotum, urethral meatus position, testicles position, genital tubercle, mullerian residues
Age of onset of genital ambiguity signs | at baseline
  years, months

CONTACTS AND LOCATIONS:
Overall Officials: Federico Baronio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (4):
- Italy (4):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - IRCCS Ospedale San Raffaele, Milan, Milano
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Pisa
  - Ospedale Pediatrico Bambino Gesù, Roma, Roma